CLINICAL TRIAL: NCT03617263
Title: Phase 2A, Double-blind, Randomized Clinical Trial to Evaluate the Efficacy and Safety of Saroglitazar Mg 4 mg Tablet Vs Placebo for Treating Nonalcoholic Fatty Liver Disease (NAFLD) in Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Saroglitazar Magnesium 4 mg in the Treatment of Nonalcoholic Fatty Liver Disease (NAFLD) in Women With PCOS (EVIDENCES VII)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SARO.17.009
Record Dates: First submitted 2018-07-23; First posted 2018-08-06 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Non-alcoholic Fatty Liver Disease in Women With PCOS
Keywords: NAFLD; PCOS; Saroglitazar Magnesium
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — saroglitazar; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Saroglitazar Magnesium 4 mg (Experimental): Saroglitazar Magnesium once daily in the morning before breakfast
  Interventions: Drug: Saroglitazar Magnesium 4 mg Tablet
- Placebo (Placebo Comparator): Placebo tablet once daily in the morning before breakfast
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saroglitazar Magnesium 4 mg Tablet — Patients randomly assigned to this group will receive Saroglitazar Magnesium orally once daily for 24 weeks.
  Other Names: Not any
  Arms: Saroglitazar Magnesium 4 mg
Drug: Placebo — Patients randomly assigned to this group will receive Placebo tablet orally once daily for 24 weeks.
  Other Names: Not any
  Arms: Placebo

SUMMARY:
This is a multicenter, phase 2A, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of Saroglitazar Magnesium in women with well characterized PCOS.

DETAILED DESCRIPTION:
This is a multicenter, phase 2A, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of Saroglitazar Magnesium in women with well characterized PCOS.

The study will be conducted over a period of up to 34 weeks and will include Screening (Days -28 to -7) Phase, a 24-week Treatment Phase following randomization on Day 1.

The primary endpoint of the study is change in hepatic fat content from baseline following 24 weeks of treatment as measured by MRI-PDFF.

ELIGIBILITY:
Inclusion Criteria:

* Females, 18 to 45 years of age.
* Previously confirmed diagnosis of PCOS:

  1. oligo-and/or anovulation;
  2. hyperandrogenism (clinical and/or biochemical);
  3. polycystic ovary morphology on ultrasonography
* Evidence of NAFLD within 6 months prior to the Screening Visit (Visit 1).
* Alanine transaminase ≥ 38 U/L at Visit 1. Visit 2 ALT must not increase >30% from Visit 1.
* Hepatic fat fraction ≥10% by MRI-PDFF.
* Willingness to participate in the study.
* Ability to understand and give informed consent for participation.
* Woman who agrees to use the contraceptive methods.

Exclusion Criteria:

* Presence of other chronic liver diseases (hepatitis B or C, autoimmune hepatitis, cholestatic liver disease, Wilsons disease, hemochromatosis, etc.).
* Average alcohol consumption ≥ 7 drinks per week for women in the 6 months prior to enrollment.
* Clinical, imaging, or histological evidence of cirrhosis.
* Patients who have used medications known to cause hepatic steatosis for more than 2 weeks in the past year.
* Prior bariatric surgery.
* Weight loss of more than 5% in the 3 months preceding screening.
* Severe co-morbidities (e.g., advanced cardiac, renal, pulmonary, or psychiatric illness).
* Known allergy, sensitivity or intolerance to Saroglitazar Magnesium, comparator or formulation ingredients.
* Use of antidiabetic and lipid lowering medications if the dose is not stable for at least the 3 months preceding screening.
* Intake of Vitamin E (>100 IU/day) or multivitamins containing Vitamin E (>100 IU/day) 3 months before enrollment.
* Use of drugs with potential effect on NAFLD/NASH in the 3 months prior to screening.
* Illicit substance abuse within the past 12 months.
* Pregnant or breast feeding females.
* Women with known Cushing syndrome or hyperprolactinemia.
* Refusal or inability to comply with the requirements of the protocol, for any reason, including scheduled clinic visits and laboratory tests.
* History of myopathies or evidence of active muscle diseases.
* History or current significant cardiovascular disease.
* History of malignancy.
* History of bladder disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deven Parmar, MD, Study Director — Zydus Therapeutics Inc.
Locations (19):
- United States (13):
  - Zydus US005, Chandler, Arizona
  - Zydus US004, Panorama City, California
  - Zydus US002, San Francisco, California
  - Zydus US008, Aurora, Colorado
  - Zydus US010, Miami, Florida
  - Zydus US001, Indianapolis, Indiana
  - Zydus US011, Morehead City, North Carolina
  - Zydus US003, Marion, Ohio
  - Zydus US015, Hershey, Pennsylvania
  - Zydus US014, Philadelphia, Pennsylvania
  - Zydus US013, Austin, Texas
  - Zydus US007, San Antonio, Texas
  - Zydus US009, San Antonio, Texas
- Mexico (6):
  - Zydus MX006, Guadalajara, Jalisco
  - Zydus MX001, Monterrey, Nuevo León
  - Zydus MX002, Monterrey, Nuevo León
  - Zydus MX005, Culiacán, Sinaloa
  - Zydus MX004, Mérida, Yucatán
  - Zydus MX003, Mexico City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelley CE, Brown AJ, Diehl AM, Setji TL. Review of nonalcoholic fatty liver disease in women with polycystic ovary syndrome. World J Gastroenterol. 2014 Oct 21;20(39):14172-84. doi: 10.3748/wjg.v20.i39.14172. PMID 25339805

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Started | 30 | 30
Completed | 26 | 26
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (7.16) | 27.2 (5.79) | 27.9 (6.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 21 | 39
  Not Hispanic or Latino | 12 | 9 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20 | 15 | 35
  Asian | 1 | 1 | 2
  Mestizo | 9 | 13 | 22
  Other | 0 | 1 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 40.14 (7.636) | 37.81 (6.981) | 38.97 (7.348)

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Fat Content
Description: Change in hepatic fat content from baseline following 24 weeks of treatment as measured by Magnetic Resonance Imaging-derived Proton Density-fat Fraction (MRI-PDFF)
Time Frame: Baseline and Week 24
Population: Per Protocol (PP) population
Measure: Least Squares Mean (Standard Error); unit: percentage of liver fat
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
percentage of liver fat | -3.1741 (1.01800) | -0.3499 (1.06137)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.0613, ANCOVA

2. Secondary Outcome: Liver Enzymes/Liver Function Tests
Description: Changes from baseline to week 12 and week 24 in Alkaline phosphatase
Time Frame: Baseline, Week 12, and Week 24
Population: Per Protocol (PP) population
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
U/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -22.64 (1.954) | -3.91 (2.083)
  Week 24 | -20.07 (2.520) | -1.66 (2.627)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p < .0001, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p < .0001, ANCOVA

3. Secondary Outcome: Liver Enzymes/Liver Function Tests
Description: Changes from baseline to week 12 and week 24 in Alanine aminotransferase
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
U/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -22.00 (4.586) | -4.72 (4.894)
  Week 24 | -25.73 (4.276) | -8.30 (4.462)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0142, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.0077, ANCOVA

4. Secondary Outcome: Liver Enzymes/Liver Function Tests
Description: Changes from baseline to week 12 and week 24 in Aspartate Aminotransferase
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
U/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -9.97 (4.233) | -3.31 (4.514)
  Week 24 | -11.27 (4.437) | -2.88 (4.627)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2893, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.1989, ANCOVA

5. Secondary Outcome: Liver Enzymes/Liver Function Tests
Description: Changes from baseline to week 12 and week 24 in gamma-glutamyl transferase
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
U/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -22.62 (2.629) | -1.52 (2.807)
  Week 24 | -21.46 (2.545) | -2.37 (2.656)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p < .0001, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p < .0001, ANCOVA

6. Secondary Outcome: Liver Enzymes/Liver Function Tests
Description: Changes from baseline to week 12 and week 24 in serum protein
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
g/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | 0.01 (0.072) | 0.02 (0.077)
  Week 24 | -0.14 (0.071) | 0.03 (0.074)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.8664, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.1137, ANCOVA

7. Secondary Outcome: Liver Enzymes/Liver Function Tests
Description: Changes from baseline to week 12 and week 24 in albumin
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
g/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | 1.06 (0.477) | -0.39 (0.510)
  Week 24 | 0.06 (0.485) | -0.15 (0.507)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0487, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.7743, ANCOVA

8. Secondary Outcome: Liver Enzymes/Liver Function Tests
Description: Changes from baseline to week 12 and week 24 in total bilirubin.
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
mg/dL
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -0.076 (0.0294) | -0.008 (0.0313)
  Week 24 | -0.066 (0.0290) | -0.004 (0.0302)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1174, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.1483, ANCOVA

9. Secondary Outcome: Insulin Resistance
Description: Evaluation of HOMA of Insulin Resistance Index determines insulin resistance and estimates insulin sensitivity, calculated by fasting insulin (μU/mL) multiplied by fasting glucose (mg/dL), and divided by a constant (405). A higher score indicates higher insulin resistance
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: Index
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
Index
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -1.983 (1.2192) | 1.081 (1.3004)
  Week 24 | 0.498 (2.1910) | 4.303 (2.2852)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0941, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.2378, ANCOVA

10. Secondary Outcome: Liver Injury
Description: Changes from baseline to week 24 in Liver Injury, including Cytokeratin (CK)-18. CK18 [M30] and CK-18 [M-65] were measured as biomarkers of hepatocyte apoptosis. Both are important indicators for liver tissue conditions and effectively reflect hepatocyte damage. A negative change from baseline indicates a decrease in hepatocyte apoptosis or a decrease in hepatocyte damage.
Time Frame: Baseline and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
U/L
  M30 | -238.801 (69.9009) | -92.160 (72.8890)
  M65 | -260.232 (100.6148) | -72.273 (104.9207)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; CK-18 Fragment - M30; Test type: Superiority; p = 0.1542, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; CK-18 Fragment - M65; Test type: Superiority; p = 0.2037, ANCOVA

11. Secondary Outcome: Liver Injury
Description: Changes from baseline to week 24 in high-sensitivity C-reactive protein (hs-CRP)
Time Frame: Baseline and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
mg/L | -1.00 (1.381) | 0.55 (1.440)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.4431, ANCOVA

12. Secondary Outcome: Liver Injury
Description: Changes from baseline to week 24 in Tumor necrosis factor (TNFα)
Time Frame: Baseline and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
ng/L | 0.109 (0.2711) | 0.587 (0.2827)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.2289, ANCOVA

13. Secondary Outcome: Liver Stiffness
Description: Changes from baseline to week 24 in liver stiffness measured by transient elastography/FibroScan
Time Frame: Baseline and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: kPa
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
kPa | -0.75 (0.953) | 1.67 (0.994)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.0853, ANCOVA

14. Secondary Outcome: Controlled Attenuation Parameter
Description: Changes from baseline to week 24 in controlled attenuation parameter measured by transient elastography/ FibroScan
Time Frame: Baseline and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: dB/m
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
dB/m | -18.84 (9.119) | -3.40 (9.521)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.2559, ANCOVA

15. Secondary Outcome: Body Mass Index (BMI)
Description: Changes from baseline to week 12 and week 24 in Body mass index
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
kg/m^2
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | 0.101 (0.2817) | 0.272 (0.3003)
  Week 24 | 0.273 (0.3132) | -0.066 (0.3266)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.6800, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.4587, ANCOVA

16. Secondary Outcome: Waist Circumference
Description: Changes from baseline to week 12 and week 24 in waist circumference
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
cm
  Week 12: number analyzed (Participants) | 25 | 21
  Week 12 | 1.285 (0.9879) | 1.142 (1.0783)
  Week 24 | 1.607 (0.8919) | 1.127 (0.9300)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.9230, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.7115, ANCOVA

17. Secondary Outcome: Changes From Baseline to Week 24 in MRI-derived Measures of Total Liver Fat Index
Description: MRI-derived measures of total liver fat index. Total liver volume: The total liver volume was calculated through a process requiring segmentation image analysis. Liver volume was calculated after complete segmentation by summing the liver surface area at each segmented slice and then multiplying this sum by individual slice thickness, in milliliters (mL). Total liver fat index: The total liver fat index (TLFI, units: % mL) took into consideration the volume of liver from which proton-density fat fraction was derived. It was calculated as the product of liver volume and the liver mean proton-density fat fraction across all liver segments.
Time Frame: Baseline and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: %mL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 22 | 23
%mL | -78.493 (38.0001) | -8.963 (37.1636)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.1983, ANCOVA

18. Secondary Outcome: Changes From Baseline to Week 24 in MRI-derived Measures of Total Liver Volume
Description: MRI-derived measures of total liver volume (Liver volume will be calculated after complete segmentation by summing the liver surface area at each segmented slice, and then multiplying this sum by individual slice thickness, in millilitres [mL])
Time Frame: Baseline and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 22 | 23
mL | -66.886 (70.3776) | -36.176 (68.8178)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.7576, ANCOVA

19. Secondary Outcome: Lipid and Lipoprotein Levels
Description: Changes from baseline to week 12 and week 24 in Triglyceride (TG)
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
mg/dL
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -41.535 (12.3535) | -21.665 (13.1733)
  Week 24 | -47.886 (15.8642) | 14.724 (16.5423)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2784, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.0091, ANCOVA

20. Secondary Outcome: Lipid and Lipoprotein Levels
Description: Changes from baseline to week 12 and week 24 in Total cholesterol (TC)
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
mg/dL
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -16.807 (3.8832) | -6.992 (4.1447)
  Week 24 | -22.650 (3.7464) | -3.120 (3.9095)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0941, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.0009, ANCOVA

21. Secondary Outcome: Lipid and Lipoprotein Levels
Description: Changes from baseline to week 12 and week 24 in High-density lipoprotein
Time Frame: Baseline, Week 12, and Week 24
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
mg/dL
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | 2.327 (1.3110) | -0.599 (1.3986)
  Week 24 | 0.676 (1.4851) | -1.561 (1.5491)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1363, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.3057, ANCOVA

22. Secondary Outcome: Lipid and Lipoprotein Levels
Description: Changes from baseline to week 12 and week 24 in Low-density lipoprotein (LDL)
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
mg/dL
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -10.318 (3.7934) | -4.821 (4.0492)
  Week 24 | -13.457 (3.0454) | -4.938 (3.1785)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3323, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.0624, ANCOVA

23. Secondary Outcome: Lipid and Lipoprotein Levels
Description: Changes from baseline to week 12 and week 24 in Small dense low density lipoprotein (sdLDL)
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
mg/dL
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -6.918 (2.0576) | -4.889 (2.1943)
  Week 24 | -9.000 (1.9510) | -2.574 (2.0346)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.5050, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.0279, ANCOVA

24. Secondary Outcome: Lipid and Lipoprotein Levels
Description: Changes from baseline to week 12 and week 24 in Very low density lipoprotein (VLDL)
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
mg/dL
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -7.102 (2.5927) | -3.521 (2.7645)
  Week 24 | -8.736 (2.9168) | 3.452 (3.0413)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3508, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.0059, ANCOVA

25. Secondary Outcome: Lipid and Lipoprotein Levels
Description: Changes from baseline apolipoprotein A
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
mg/dL
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | 4.486 (3.8760) | 2.130 (4.1326)
  Week 24 | -2.830 (3.1112) | -1.272 (3.2442)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.6800, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.7310, ANCOVA

26. Secondary Outcome: Lipid and Lipoprotein Levels
Description: Changes from baseline in apolipoprotein B
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
mg/dL
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -10.673 (2.7834) | -3.508 (2.9723)
  Week 24 | -13.146 (2.3060) | -3.233 (2.4071)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0896, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.0053, ANCOVA

27. Secondary Outcome: Sex Hormone Binding Globulin (SHBG) Level
Description: Changes from baseline in SHBG level
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
nmol/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | 17.182 (13.1496) | 27.506 (14.0281)
  Week 24 | -3.882 (8.0521) | 8.286 (8.3982)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.5962, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.3035, ANCOVA

28. Secondary Outcome: Ovarian Function
Description: Changes from baseline in 17-hydroxyprogesterone
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: ng/dL
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
ng/dL
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | 8.800 (9.7348) | -4.819 (10.3892)
  Week 24 | -10.325 (6.8372) | -2.168 (7.1337)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3482, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.4176, ANCOVA

29. Secondary Outcome: Ovarian Function
Description: Changes from baseline in Total testosterone
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
nmol/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -0.173 (0.1134) | -0.171 (0.1209)
  Week 24 | -0.231 (0.1182) | -0.073 (0.1233)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.9930, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.3612, ANCOVA

30. Secondary Outcome: Ovarian Function
Description: Changes from baseline in free testosterone
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
nmol/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -0.005 (0.0028) | -0.009 (0.0030)
  Week 24 | -0.005 (0.0028) | -0.003 (0.0029)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4373, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.6248, ANCOVA

31. Secondary Outcome: Ovarian Function
Description: Changes from baseline in follicle-stimulating hormone (FSH)
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
IU/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -0.892 (0.3356) | -1.722 (0.3580)
  Week 24 | -0.689 (0.3196) | -1.125 (0.3334)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0994, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.3527, ANCOVA

32. Secondary Outcome: Ovarian Function
Description: Changes from baseline in luteinizing hormone (LH)
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
IU/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -1.140 (0.8881) | -1.632 (0.9467)
  Week 24 | -1.305 (1.2020) | 0.140 (1.2532)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.7065, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.4096, ANCOVA

33. Secondary Outcome: Ovarian Function
Description: Changes from baseline in LH-to-FSH ratio
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 24 | 22
Ratio
  Week 12 | -0.230 (0.1731) | 0.064 (0.1808)
  Week 24 | -0.324 (0.2226) | 0.136 (0.2326)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2475, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.1621, ANCOVA

34. Secondary Outcome: Ovarian Function
Description: Changes from baseline in estradiol
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
pmol/L
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -57.237 (41.4020) | -24.045 (44.1354)
  Week 24 | -105.380 (65.5983) | 17.209 (68.3930)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.5862, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.2026, ANCOVA

35. Secondary Outcome: Changes From Baseline to Week 12 and Week 24 in Free Androgen Index
Description: Free androgen index is a ratio used to determine abnormal androgen status in humans, measured by Total testosterone level divided by the sex hormone binding globulin (SHBG) level, and then multiplying by a constant, usually 100. A higher score indicates a worse outcome (more androgenic).
Time Frame: Baseline, Week 12, and Week 24
Population: PP population
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23
Ratio
  Week 12: number analyzed (Participants) | 25 | 22
  Week 12 | -0.371 (0.1637) | -0.483 (0.1746)
  Week 24 | -0.253 (0.1742) | -0.256 (0.1816)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 12; Test type: Superiority; p = 0.6434, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Week 24; Test type: Superiority; p = 0.9895, ANCOVA

36. Secondary Outcome: Peak Plasma Concentration [Cmax] (For Single Dose)
Description: Pharmacokinetics of Saroglitazar following first dose
Time Frame: PK sampling timepoints: pre-dose (0.0), 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, and 24 hours post-dose of First dose (visit 3)
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 10
ng/mL | 120.250 (49.997)

37. Secondary Outcome: Time to Reach Peak Plasma Concentration [Tmax] (For Single Dose)
Description: Pharmacokinetics of Saroglitazar following first dose
Time Frame: as for outcome 36
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 10
hour | 1.902 (1.103)

38. Secondary Outcome: Area Under Plasma Concentration vs. Time Curve Till the Last Time Point [AUC0-t] (For Single Dose)
Description: Pharmacokinetics of Saroglitazar following first dose
Time Frame: as for outcome 36
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 10
ng*hr/mL | 486.033 (188.320)

39. Secondary Outcome: Area Under Plasma Concentration vs. Time Curve Extrapolated to the Infinity (AUC0-∞) After First Dose (For Single Dose)
Description: Pharmacokinetics of Saroglitazar following first dose
Time Frame: as for outcome 36
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 10
ng/mL*hr | 473.771 (182.430)

40. Secondary Outcome: Area Under Plasma Concentration vs. Time Curve in a 24 h Dosing Interval (AUCtau) After First Dose (For Single Dose)
Description: Pharmacokinetics of Saroglitazar following first dose
Time Frame: as for outcome 36
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 10
ng*hr/mL | 491.981 (192.373)

41. Secondary Outcome: Elimination Rate Constant [Kel] (For Single Dose)
Description: Pharmacokinetics of Saroglitazar following first dose
Time Frame: as for outcome 36
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 10
1/hr | 0.144 (0.057)

42. Secondary Outcome: Elimination Half-life [tHalf] (For Single Dose)
Description: Pharmacokinetics of Saroglitazar following first dose
Time Frame: as for outcome 36
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 10
hr | 5.317 (1.559)

43. Secondary Outcome: Apparent Volume of Distribution [Vd/F] (For Single Dose)
Description: Pharmacokinetics of Saroglitazar following first dose
Time Frame: as for outcome 36
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 10
L | 77.890 (42.887)

44. Secondary Outcome: Apparent Clearance [CL/F] (For Single Dose)
Description: Pharmacokinetics of Saroglitazar following first dose
Time Frame: as for outcome 36
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 10
L/hr | 9.305 (3.599)

45. Secondary Outcome: Peak Plasma Concentration [Cmax,ss] (For Multiple Dose)
Description: Pharmacokinetics of Saroglitazar following last dose
Time Frame: PK sampling timepoints: pre-dose (0.0), 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0,10.0, and 24 hours post-dose of Last dose (Visit 8)
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 9
ng/mL | 137.210 (57.770)

46. Secondary Outcome: Time to Reach Peak Plasma Concentration [Tmax,ss] (For Multiple Dose)
Description: Pharmacokinetics of Saroglitazar following last dose
Time Frame: PK sampling timepoints: pre-dose (0.0), 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, and 24 hours post-dose of Last dose (visit 8)
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 9
hour | 1.667 (0.866)

47. Secondary Outcome: Area Under Plasma Concentration vs. Time Curve in a 24 h Dosing Interval (AUCtau) After Last Dose (For Multiple Dose)
Description: Pharmacokinetics of Saroglitazar following last dose
Time Frame: as for outcome 46
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 9
ng*hr/mL | 454.916 (162.275)

48. Secondary Outcome: Elimination Rate Constant [Kel,ss] (For Multiple Dose)
Description: Pharmacokinetics of Saroglitazar following last dose
Time Frame: as for outcome 46
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 9
1/hr | 0.147 (0.047)

49. Secondary Outcome: Elimination Half-life [Thalf,ss] (For Multiple Dose)
Description: Pharmacokinetics of Saroglitazar following last dose
Time Frame: as for outcome 46
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 9
hour | 5.196 (1.790)

50. Secondary Outcome: Apparent Volume of Distribution [Vd/F,ss] (For Multiple Dose)
Description: Pharmacokinetics of Saroglitazar following last dose
Time Frame: as for outcome 46
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 9
L | 66.047 (28.325)

51. Secondary Outcome: Apparent Clearance [CL/F,ss] (For Multiple Dose)
Description: Pharmacokinetics of Saroglitazar following last dose
Time Frame: as for outcome 46
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 9
L/hr | 8.883 (2.444)

52. Secondary Outcome: Minimal or Trough Plasma Concentration [Cmin] (For Multiple Dose)
Description: Pharmacokinetics of Saroglitazar following last dose
Time Frame: as for outcome 46
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 9
ng/mL | 1.053 (0.825)

53. Secondary Outcome: Fluctuation Index (For Multiple Dose)
Description: Pharmacokinetics of Saroglitazar following the last dose. It is calculated as (Cmax - Cmin) / Cavg. The value has been multiplied by 100, hence has been expressed in percentage unit; where Cmax is the Maximum measured plasma concentration at steady state, Cmin is Minimal or trough plasma concentration at steady state, and Cavg is Average concentration = AUCtau,ss /tau.
Time Frame: as for outcome 46
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 9
percentage | 676.702 (240.892)

54. Secondary Outcome: Accumulation Index Calculated as a Ratio of AUCtau (Last Dose)/AUCtau (First Dose) (For Multiple Dose)
Description: Pharmacokinetics of Saroglitazar following last dose
Time Frame: as for outcome 46
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 9
ratio | 1.113 (0.264)

ADVERSE EVENTS:
Time Frame: 30 weeks
Description: Treatment-emergent adverse events (TEAEs)
Arm/Group | Saroglitazar Magnesium 4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 19/30 | 22/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saroglitazar Magnesium 4 mg (N=30) | Placebo (N=30)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Covid-19 (Infections and infestations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (8) | 1 (1)
General disorders and administration site conditions (General disorders) | 3 (3) | 4 (5)
Dysmenorrhea (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
ALT increased (Investigations) | 0 (0) | 2 (2)
AST increased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT03617263/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT03617263/SAP_001.pdf